CLINICAL TRIAL: NCT06216678
Title: The Effects of Healthy Diets With Plant Oils on Heart and Metabolic Health: A Randomized, Crossover, Controlled-feeding Study
Brief Title: The Effects of Healthy Diets With Plant Oils on Heart and Metabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Cotton Incorporated (Unknown)
Responsible Party: Principal Investigator, Kristina Petersen PhD, APD, FAHA, Associate Professor, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: POS
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Cottonseed Oil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Diet + Cottonseed Oil (CSOD) (Experimental): Healthy dietary pattern containing 40g/day/2000 kcal of cottonseed oil (CSO)
  Interventions: Other: Healthy Dietary Pattern with Cottonseed Oil
- Healthy Diet + Fatty Acid-Matched Plant Oils (FAMD) (Active Comparator): Healthy dietary pattern containing 40g/day/2000 kcal of a blend of plant oils comprising a fatty acid profile that matches the CSOD but devoid of CSO
  Interventions: Other: Healthy Dietary Pattern with Fatty Acid-Matched Plant Oils
- Healthy Diet + PUFA:SFA Ratio-Matched Plant Oil (P:S-MD) (Active Comparator): Healthy dietary pattern containing 40g/day/2000 kcal of plant oil that is lower in polyunsaturated fatty acids (PUFA) and saturated fatty acids (SFA) than the CSOD, but with a matched PUFA:SFA ratio and devoid of CSO.
  Interventions: Other: Healthy Dietary Pattern with PUFA:SFA Ratio-Matched Plant Oil

INTERVENTIONS:
Other: Healthy Dietary Pattern with Cottonseed Oil — Cottonseed Oil
  Arms: Healthy Diet + Cottonseed Oil (CSOD)
Other: Healthy Dietary Pattern with Fatty Acid-Matched Plant Oils — Plant oil blend fatty acid matched
  Arms: Healthy Diet + Fatty Acid-Matched Plant Oils (FAMD)
Other: Healthy Dietary Pattern with PUFA:SFA Ratio-Matched Plant Oil — Plant oil with matched PUFA to SFA ratio
  Arms: Healthy Diet + PUFA:SFA Ratio-Matched Plant Oil (P:S-MD)

SUMMARY:
This study will examine the effect of a healthy diet containing cottonseed oil compared to healthy diets containing other commonly consumed plant oils on biomarkers of heart and metabolic health after 4 weeks.

DETAILED DESCRIPTION:
This is a 3-period randomized crossover complete feeding study examining if a dietary pattern containing cottonseed oil improves lipids/lipoproteins and other cardiometabolic disease risk factors to a greater extent than a fatty acid matched diet devoid of cottonseed oil and a diet lower in polyunsaturated fatty acids (PUFA) and saturated fatty acids (SFA), but with a matched PUFA:SFA ratio

ELIGIBILITY:
Inclusion Criteria:

* LDL-C ≥100 mg/dL and ≤190 mg/dL
* BMI of 25-40 kg/m2
* Blood pressure <140/90 mmHg
* Fasting blood glucose <126 mg/dL
* Fasting triglycerides <350 mg/dL
* ≤10% change in body weight for 6 months prior to enrollment

Exclusion Criteria:

* Type 1 or type 2 diabetes or fasting blood glucose ≥126 mg/dL
* Prescription of anti-hypertensive, lipid lowering or glucose lowering drugs
* Intake of supplements that affect the outcomes of interest and unwilling to cease during the study period
* Diagnosed liver, kidney, or autoimmune disease
* Prior cardiovascular event (e.g., stroke, heart attack)
* Current pregnancy or intention of pregnancy within the next 6 months
* Lactation within prior 6 months
* Follows a vegetarian or vegan diet
* Food allergies/intolerance/sensitives/dislikes of foods included in the study menu
* Antibiotic use within the prior 1 month
* Oral steroid use within the prior 1 month
* Use of tobacco or nicotine containing products with in the past 6 months
* Cancer any site within the past 10 years (eligible if ≥10 years without recurrence) or non-melanoma skin cancer with in the past 5 years (eligible if ≥5 years without recurrence)
* Participation in another clinical trial within 30 days of baseline
* Currently following a restricted or weight loss diet
* Prior bariatric surgery
* Intake of >14 alcoholic drinks/week and/or lack of willingness to consume a maximum of two standard drinks per week while enrolled in the study and/or not willing to avoid alcohol consumption for 48 hour prior to test visits

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
LDL-cholesterol concentration | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL. LDL-cholesterol will be measured directly via enzymatic assay. The mean of the LDL-cholesterol values from day 1 and day 2 testing will be used for analysis.

SECONDARY OUTCOMES:
Triglycerides concentration | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL
Total Cholesterol concentration | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL
HDL-cholesterol concentration | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL
Particle Size and Number of LDL, HDL, VLDL and Chylomicrons | 4 weeks
  Measured via Nuclear Magnetic Resonance
Central Systolic and Diastolic Blood Pressure | 4 weeks
  Blood pressure measured assessed using a SphymoCor Xcel (Atcor Medical)
Brachial Systolic and Diastolic Blood Pressure | 4 weeks
  Blood pressure measured assessed using a SphymoCor Xcel (Atcor Medical)
Carotid-Femoral Pulse Wave Velocity | 4 weeks
  A measure of arterial stiffness assessed using a SphymoCor Xcel (Atcor Medical).
  Expressed in meters/second.
Fasting Serum Insulin concentration | 4 weeks
  Serum insulin levels assessed in a fasting blood draw and expressed in micro IU/mL
Fasting Plasma Glucose concentration | 4 weeks
  Glucose assessed in a fasting blood draw and expressed in mg/dL
Fasting Serum Fructosamine concentration | 4 weeks
  Fructosamine assessed in a fasting blood draw and expressed in micro IU/mL
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 4 weeks
  Calculated from insulin and glucose measured from a fasting blood sample. Calculated as (insulin × glucose) / 22.5
Dihydrosterculic acid | 4 weeks
  Dihydrosterculic acid assessed from fasting blood draw and measured using Gas-Chromatography-Mass Spectrometry

OTHER OUTCOMES:
Composition of the Gut Microbiota | 4 weeks
  Abundance measured using 16 s rRNA sequencing
Fatty acids | 4 weeks
  Fatty acid analysis of red blood cells assessed from fasting blood draw and measured using Gas Chromatography

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be deposited into an open access repository once results from all pre-specified primary and secondary outcomes are published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication of all pre-specified primary and secondary outcomes

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT06216678/SAP_001.pdf